CLINICAL TRIAL: NCT01387269
Title: Anamorelin HCl in the Treatment of Non-Small Cell Lung Cancer-Cachexia (NSCLC-C): A Randomized Double-Blind Placebo-Controlled Multicenter Phase III Study to Evaluate the Safety and Efficacy of Anamorelin HCl in Patients With NSCLC-C
Brief Title: Safety and Efficacy of Anamorelin HCl in Patients With Non-Small Cell Lung Cancer-Cachexia (ROMANA 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT-ANAM-301
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Cachexia; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Cachexia; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 mg QD (Experimental): Anamorelin HCL 100 mg will be administered daily
  Interventions: Drug: Anamorelin HCl
- Placebo (Placebo Comparator): Placebo tablets identical in appearance to active tablets; oral administration once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anamorelin HCl — Anamorelin HCl will be orally administered daily at least one hour before meal
  Arms: 100 mg QD
Drug: Placebo — Placebo tablets identical in appearance to active tablets; oral administration QD for 12 weeks, at least 1 hour before meal
  Arms: Placebo

SUMMARY:
The administration of Anamorelin in patients with Stage III-IV non-small cell lung cancer-cachexia (NSCLC-C) is expected to increase appetite, lean body mass, weight gain, and muscle strength.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter study to assess the safety and efficacy of Anamorelin in patients with non-small cell lung cancer-cachexia (NSCLC-C). The primary efficacy analysis will include the treatment difference in the change in lean body mass and physical function. Pharmacokinetic (PK) samples will also be collected at Day 43 visit for population PK.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of unresectable Stage III or Stage IV NSCLC
* Patients may be receiving maintenance chemotherapy
* Patients planning to initiate a new chemotherapy and/or radiation therapy regimen may do so only within ± 14 days of randomization
* Patients may have completed a chemotherapy and/or radiation therapy and/or have no plan to initiate a new regimen within 12 weeks from randomization; at least 14 days must elapse from the completion of the chemotherapy and/or radiation therapy prior to randomization
* Involuntary weight loss of ≥5% body weight within 6 months prior to screening or a screening body mass index (BMI) <20 kg/m2
* Body mass index ≤30 kg/m2
* Life expectancy of >4 months at time of screening
* ECOG performance status ≤2
* Adequate hepatic function, defined as AST and ALT levels ≤5 x upper limit of normal
* Adequate renal function, defined as creatinine ≤2 x upper limit of normal, or calculated creatinine clearance >30 ml/minute
* Ability to understand and comply with the procedures for the HGS evaluation
* If a woman of childbearing potential or a fertile man, he/she must agree to use an effective form of contraception during the study and for 30 days following the last dose of study drug (an effective form of contraception is abstinence, a hormonal contraceptive, or a double-barrier method)
* Must be willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the protocol tests and procedures

Exclusion Criteria:

* Other forms of lung cancer (e.g., small cell, mesothelioma)
* Women who are pregnant or breast-feeding
* Known HIV, hepatitis (B&C), or active tuberculosis
* Had major surgery (central venous access placement and tumor biopsies are not considered major surgery) within 4 weeks prior to randomization; patients must be well recovered from acute effects of surgery prior to screening; patients should not have plans to undergo major surgical procedures during the treatment period
* Currently taking prescription medications intended to increase appetite or treat weight loss; these include, but are not limited to, testosterone, androgenic compounds, megestrol acetate, methylphenidate, and dronabinol
* Inability to readily swallow oral tablets; patients with severe gastrointestinal disease (including esophagitis, gastritis, malabsorption, or obstructive symptoms) or intractable or frequent vomiting are excluded
* Has an active, uncontrolled infection
* Has uncontrolled diabetes mellitus
* Has untreated clinically relevant hypothyroidism
* Has known or symptomatic brain metastases
* Receiving strong CYP3A4 inhibitors within 14 days of randomization
* Receiving tube feedings or parenteral nutrition (either total or partial); patients must have discontinued these treatments for at least 6 weeks prior to Day 1, and throughout the study duration
* Other clinical diagnosis, ongoing or intercurrent illness that in the Investigator's opinion would prevent the patient's participation
* Has had previous exposure to Anamorelin HCl
* Patients actively receiving a concurrent investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (12):
  - Fullerton, California
  - Glendale, California
  - La Jolla, California
  - Riverside, California
  - Orange City, Florida
  - Quincy, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Northport, New York
  - Cincinnati, Ohio
  - Houston, Texas
- Belarus (3):
  - Brest
  - Lesnoy
  - Minsk
- Belgium (4):
  - Antwerp
  - Brussels
  - Genk
  - Liège
- Canada (4):
  - Edmonton, Alberta
  - Sault Ste. Marie, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (5):
  - Benešov
  - Brno
  - Hlučín
  - Liberec
  - Nymburk
- France (2):
  - Lyon
  - Villejuif
- Germany (4):
  - Berlin
  - Großhansdorf
  - Halle
  - Minden
- Budapest, Hungary
- Italy (2):
  - Placenza
  - Rozzano
- Netherlands (4):
  - Amsterdam
  - Goes
  - Maastricht
  - Nieuwegein
- Poland (4):
  - Grudziądz
  - Katowice
  - Krakow
  - Lublin
- Russia (2):
  - Saint Petersburg
  - Yekaterinburg
- Serbia (2):
  - Belgrade
  - Kamenitz
- Slovenia (2):
  - Golnik
  - Ljubljana
- Spain (4):
  - Barcelona
  - Córdoba
  - Seville
  - Valencia
- Ukraine (5):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kyiv
  - Zaporizhzhya

REFERENCES:
- [Derived] Laird BJA, Skipworth R, Bonomi PD, Fallon M, Kaasa S, Giorgino R, McMillan DC, Currow DC. Anamorelin Efficacy in Non-Small-Cell Lung Cancer Patients With Cachexia: Insights From ROMANA 1 and ROMANA 2. J Cachexia Sarcopenia Muscle. 2025 Feb;16(1):e13732. doi: 10.1002/jcsm.13732. PMID 39992021
- [Derived] Currow D, Temel JS, Abernethy A, Milanowski J, Friend J, Fearon KC. ROMANA 3: a phase 3 safety extension study of anamorelin in advanced non-small-cell lung cancer (NSCLC) patients with cachexia. Ann Oncol. 2017 Aug 1;28(8):1949-1956. doi: 10.1093/annonc/mdx192. PMID 28472437
- [Derived] Temel JS, Abernethy AP, Currow DC, Friend J, Duus EM, Yan Y, Fearon KC. Anamorelin in patients with non-small-cell lung cancer and cachexia (ROMANA 1 and ROMANA 2): results from two randomised, double-blind, phase 3 trials. Lancet Oncol. 2016 Apr;17(4):519-531. doi: 10.1016/S1470-2045(15)00558-6. Epub 2016 Feb 20. PMID 26906526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 477 patients with advanced NSCLC-C (defined as unresectable Stage III and Stage IV and a weight loss of ≥ 5% body weight within 6 months prior to screening or a screening body mass index [BMI] < 20 kg/m2) were to be randomized 2:1 to anamorelin HCl 100 mg or placebo.
Pre-assignment Details: Central randomization stratified patients by geographic region, by chemotherapy and/or radiation therapy status and by weight loss over prior 6 months.
Groups:
- Anamorelin HCl: Active drug; 100 mg tablets; oral administration QD for 12 weeks, at least 1 hour before the first meal of the day.
- Placebo: Placebo tablets identical in appearance to active tablets; oral administration QD for 12 weeks, at least 1 hour before the first meal of the day.
Period: Overall Study
Arm/Group | Anamorelin HCl | Placebo
Started | 323 | 161
ITT Population | 323 | 161
MITT Population | 284 | 141
Safety Population | 320 | 161
Completed (A patient was considered to have completed the study if the patient completed Week 12/Day 85 Visit.) | 231 | 121
Not Completed | 92 | 40
Not completed — Death | 38 | 20
Not completed — Other | 8 | 7
Not completed — Unrelated AE | 12 | 3
Not completed — Withdrawal by patient | 32 | 10
Not completed — Study drug-related AE | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) Population included all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anamorelin HCl | Placebo | Total
Number analyzed (Participants) | 323 | 161 | 484
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 215 | 105 | 320
  >=65 years | 108 | 56 | 164
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 40 | 116
  Male | 247 | 121 | 368
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 319 | 159 | 478
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Russian Federation | 8 | 4 | 12
  Serbia | 10 | 3 | 13
  Ukraine | 133 | 66 | 199
  Belarus | 15 | 9 | 24
  United States | 26 | 11 | 37
  Canada | 9 | 6 | 15
  Netherlands | 2 | 0 | 2
  Poland | 48 | 26 | 74
  Slovenia | 5 | 4 | 9
  Spain | 13 | 3 | 16
  Belgium | 11 | 4 | 15
  Czech Republic | 16 | 11 | 27
  France | 8 | 6 | 14
  Germany | 10 | 3 | 13
  Italy | 9 | 5 | 14
Geographic region [Count of Participants; unit: Participants]
  North America | 35 | 17 | 52
  West Europe | 122 | 62 | 184
  East Europe + Russia | 166 | 82 | 248
  Australia | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Lean Body Mass
Description: Change in Lean Body Mass (LBM) from baseline over 12 weeks for the ITT Population. Change from baseline over 12 weeks was defined as the average of the change from baseline at Week 6 and the change from baseline at Week 12.
Time Frame: Change in Lean Body Mass from Baseline Over 12 Weeks
Population: Intent-to-Treat Population. Some patients in the ITT population were excluded from the primary LBM/HGS analysis (i.e., multiple imputations/ranking method) if they survived to Week 12 but missed their baseline covariates including LBM, HGS, or ECOG OR had Week 6 and Week 12 outcomes that were outside the visit windows.
Measure: Median (95% Confidence Interval); unit: kg
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 316 | 158
kg | 0.99 [0.61 to 1.36] | -0.47 [-1.00 to 0.21]
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank sum test

2. Primary Outcome: Change in Handgrip Strength
Description: Change in Handgrip Strength (HGS) of the non-dominant hand from baseline over 12 weeks for the ITT Population. Change from baseline over 12 weeks was defined as the average of the change from baseline at Week 6 and the change from baseline at Week 12.
Time Frame: Change in Handgrip Strength of the Non-Dominant Hand from Baseline Over 12 Weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: kg
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 316 | 158
kg | -1.10 [-1.69 to -0.40] | -1.58 [-2.99 to -1.14]
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p = 0.1475, Wilcoxon rank sum test

3. Secondary Outcome: Change in A/CS Domain Score
Description: The Functional Assessment of Anorexia/Cachexia Treatment (FAACT) Additional Concerns Subscale (A/CS domain) is a 12-item scale that is part of the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System. Each item is answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).
  The 12-items are summed together to obtain the domain score. Note that negatively phrased questions are reverse scored so that higher scores always represent improvement/less symptom burden. The total possible score for the A/CS domain ranges from 0 (worst) to 48 (best).
Time Frame: Change in FAACT A/CS Domain Score from Baseline Over 12 Weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 284 | 141
scores on a scale | 4.12 (0.752) | 1.92 (0.805)
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis

4. Secondary Outcome: Change in FACIT-F Fatigue Domain Score
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) fatigue domain is a 13-item scale that is part of the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System. Each item is answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).
  The 13-items are summed together to obtain the domain score. Note that negatively phrased questions are reverse scored so that higher scores always represent improvement/less symptom burden. The total possible score for the FACIT-F fatigue domain ranges from 0 (worst) to 52 (best).
Time Frame: Change in FACIT-F Fatigue Domain Score from Baseline Over 12 Weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 284 | 141
scores on a scale | 0.26 (0.886) | -1.19 (0.933)
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p = 0.0544, Mixed Models Analysis

5. Secondary Outcome: Change in Body Weight
Description: Change in body weight (BW) from baseline overall (i.e., over 12 weeks) for the MITT Population.
Time Frame: Change in Body Weight from Baseline Over 12 Weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Anamorelin HCl | Placebo
Number analyzed (Participants) | 284 | 141
kg | 2.20 (0.326) | 0.14 (0.363)
Statistical Analysis 1: Comparison: Anamorelin HCl vs Placebo; Superiority analysis; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events that occurred during the clinical trial, commenced with the first dose of study drug through the 28 day post-treatment follow-up visit.
Description: Adverse events that occurred following the signature of the informed consent, but prior to the first dose of study drug were not reported as adverse events in this trial. The adverse event reporting period also ended if the patient began an alternative therapy within 28 days of the last administration of study drug. The Safety Population, defined as all randomized patients who received any study drug, was used for all safety analyses.
Arm/Group | Anamorelin HCl | Placebo
Serious Adverse Events (participants affected / at risk) | 82/320 | 48/161
Other Adverse Events (participants affected / at risk) | 182/320 | 84/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin HCl (N=320) | Placebo (N=161)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Inferior vena caval occlusion (Vascular disorders) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 (24) | 12 (12)
Death (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 4 (5)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin HCl (N=320) | Placebo (N=161)
Alanine aminotransferase increased (Investigations) | 50 (78) | 14 (20)
Aspartate aminotransferase increased (Investigations) | 37 (52) | 15 (21)
Blood alkaline phosphatase increased (Investigations) | 34 (40) | 10 (14)
Platelet count decreased (Investigations) | 14 (30) | 10 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (24) | 11 (13)
Anaemia (Blood and lymphatic system disorders) | 119 (179) | 66 (114)
Leukopenia (Blood and lymphatic system disorders) | 16 (17) | 10 (10)
Neutropenia (Blood and lymphatic system disorders) | 28 (34) | 22 (34)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (42) | 23 (34)
Asthenia (General disorders) | 19 (23) | 9 (10)
Fatigue (General disorders) | 25 (28) | 13 (15)
Pyrexia (General disorders) | 15 (16) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 17 (21) | 9 (9)
Nausea (Gastrointestinal disorders) | 29 (44) | 15 (21)
Vomiting (Gastrointestinal disorders) | 25 (27) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 13 (15) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 35 (41) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor intends to publish the complete study results in a timely manner that is appropriate to the project. Separate publication of a portion of the study results by any PI is discouraged.